CLINICAL TRIAL: NCT04071145
Title: Using Sensors to Measure Drug Concentrations in Exhaled Breath
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nadav Goldental (Other)
Responsible Party: Sponsor-Investigator, Nadav Goldental, Principal investigator, The Chaim Sheba Medical Center
Organization: The Chaim Sheba Medical Center (Other)
Other Study IDs: 6419-19-SMC
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of blood tests to measure drug concentrations in psychiatric patients is often a crucial part of monitoring and evaluating the course of treatment. Such tests are commonly conducted as part of official protocols, and patients are often tested on a weekly basis.

The current study aims to examine the possibility of using a novel, non-invasive device to measure drug concentrations in exhaled breath as an alternative to blood tests. The device, SniffPhone, uses sensors to detect and measure volatile organic compounds (VOCs) in exhaled breath, and features a small and portable design. Sniff Phone has been previously approved for use in clinical trials and has been used successfully to screen for particular types of cancer and other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Proper ability to give informed consent
* Psychiatric patients undergoing treatment at Sheba Medical Center
* Patients with treatment plans that require therapeutic drug monitoring

Exclusion Criteria:

* Involuntary psychiatric hospitalization
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients with traetment plans that require theraputic drug monitoring
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Detection of drug type and concentration in volatile organic compounds (VOCs) profile | Up to 6 months
  Detection of drug type and concentration in VOCs profile (measured using Sniff Phone)
Correlation between drug concentration and volatile organic compounds VOC concentrations | Up to 6 months
  Correlation between drug concentration (as measured in blood test) and VOCs (hexanone acetic acid, heptane, hexanal, 3-heptanone, hexanoic acid, heptanal and nonanal) measured using Sniff Phone.